CLINICAL TRIAL: NCT00428805
Title: Site Specific Approaches to Prevention or Management of Pediatric Obesity: Child Health Initiative for Lifelong Eating and Exercise--CHILE
Brief Title: Child Health Initiative for Lifelong Eating and Exercise (CHILE)
Acronym: CHILE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Based on the primary study completion date, this research does not meet the former definition of a clinical trial.
Sponsor: University of New Mexico (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sally Davis, principal investigator, University of New Mexico
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: DK72958; R01DK072958 (NIH)
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Obesity
Keywords: body composition; physical activity; dietary intake; children
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention 1 (Experimental): This transcommunity study has one intervention and one control group. The intervention, described elsewhere has 6 components--classroom curriculum, family component,grocery store component, health care provider component, training for Head Start food service workers,and training for Head Start teachers/aides.
  Interventions: Behavioral: classroom curriculum; Behavioral: In-service training for Head Start teachers/aides; Behavioral: Training for Head Start food service; Behavioral: Family intervention component; Behavioral: Food source; Behavioral: Health care providers; Behavioral: CHILE Head Start Intervention
- control 2 (No Intervention): measurement only control arm

INTERVENTIONS:
Behavioral: classroom curriculum — classroom curriculum for 3 & 4 year old children includes activities to increase intake of fruits, vegetables, & whole grains; increase physical activity; decrease intake of fats and sugared drinks; and decrease screen time following monthly learning modules.
  Teachers are trained to carry out the classroom curriculum.
  Arms: intervention 1
Behavioral: In-service training for Head Start teachers/aides — Teachers and teacher aides are trained quarterly by certified trainers and receive a certificate for participating in the training. Topics include the content as well as developmental concepts.
  Arms: intervention 1
Behavioral: Training for Head Start food service — Food service workers are trained (quarterly) to modify food ordering, food preparation, and food serving to match the aims of the study
  Arms: intervention 1
Behavioral: Family intervention component — Families receive the CHILE intervention quarterly at Family Events. These include family activities to increase intake of fruits, vegetables, whole grains, decrease intake of fats and sugared drinks, increase of physical activity and decrease screen time. Parenting skills are also included.
  Arms: intervention 1
Behavioral: Food source — The grocery store component includes field trips, self labeling, and taste testing of promoted foods.
  Arms: intervention 1
Behavioral: Health care providers — The health care provider component includes the health care providers presenting at the Family Events and reinforcing the CHILE intervention message in the practice setting when talking with families of head start children.
  Arms: intervention 1
Behavioral: CHILE Head Start Intervention — There are six components of this transcommunity social-ecological intervention including a classroom curriculum, health care provider component, family component, training of Head Start teachers/aides, training of food service staff and grocery store component.
  Arms: intervention 1

SUMMARY:
Child Health Initiative for Lifelong Eating and Exercise (CHILE) is a trans-community multidisciplinary site-specific intervention and evaluation plan for a Head Start and family-based culturally and developmentally appropriate intervention. The primary goals are to increase physical activity and improve dietary intake through increased consumption of fruits, vegetables and whole grain and decrease consumption of sweetened drinks and high-fat foods,decrease television and other screen time, and decrease obesity in three to five year old Hispanic and American Indian children enrolled in Head Start programs in rural New Mexico. The trans-community intervention includes: A classroom curriculum for children; an in-service training program for Head Start teachers and educational aides; a school food service component; a family intervention; a community leader/local health care provider component; and a grocery store component.

Participants include 16 Head Start programs serving Hispanic and Native American children and families from underserved communities in rural New Mexico. This is a randomized trial with an Intervention Condition and Control Condition. One cohort of three-year old Head Start students will be followed and measured for two years. During the two years in Head Start those children, their teachers, and families enrolled in the Intervention Condition will receive a program of activities to modify their dietary, physical activity, and screen viewing behaviors. Also addressed are the Head Start and community environments and policies, local grocery stores, and health care providers.

CHILE uses an ecological framework including social cognitive theory, intervention mapping, environmental and policy changes, developmental theory, and sound educational practices. The approach includes in from the community to ensure acceptability, cultural appropriateness, feasibility, sustainability, and later transferability to similar communities.

The primary outcome measures include changes in physical activity levels, dietary fiber intake, dietary fat intake, intake of sugared drinks, television viewing and other screen time, in BMI. Secondary measures include changes in the Head Start and community environments and policies related to physical activity, school food service, school snacks, and availability of healthful options. We will also examine the role of community leaders, especially health care providers, in raising awareness and creating a supportive and sustainable environment for the prevention of obesity.

DETAILED DESCRIPTION:
The purpose of this study is to design, implement, and evaluate a culturally appropriate, multi-level trans-community obesity prevention for Head Start staff, children, and their families in rural American Indian and Hispanic communities in New Mexico. The intervention, Child Health Initiative for Lifelong Eating and Exercise (CHILE) includes policy changes to address environmental determinants of healthful eating and physical activity behaviors, as well as individual and interpersonal level strategies to influence behavioral determinants. CHILE will promote increased moderate to vigorous physical activity; increased consumption of fruits, vegetables, and whole grains; decreased consumption of sweetened beverages and high-fat foods; and decreased television viewing and other screen time.

This study will employ a nested design in which 16 Head Start programs are randomly assigned to the intervention (n=8) or the control condition (n=8). Two cohorts of 3-year-old children within each Head Start center will be followed for two years post randomization. Participants will be assessed using a measurement interview protocol a total of four times: pre-intervention, twice during intervention, and two years post intervention. One of the midpoint time points will collect height and weight measurements only. This longitudinal component of the design will allow for an in-depth understanding of the processes at work in the intervention and an exploration of the hypothesized mediating effects, as well as potential moderators, such as individual characteristics of participants that may influence intervention exposure or efficacy. In order to more efficiently address these goals, the study has been divided into three phases.

Phase I will take place over the first 16 months of the study. During this time the focus will be on the identification and recruitment of Head Start centers, formative assessment with all Head Start centers, randomization of Head Start centers to the intervention or control condition, obtaining institutional review board approvals, intervention planning with intervention Head Start centers and their communities, and preparation and pilot testing of the measurement protocols.

Sixteen rural Head Start centers in predominately American Indian (6 centers) and Hispanic (10 centers) communities in NM are being recruited with the assistance of our community partners and through site visits, phone calls, and letters. In order to participate in this study, the Head Start Director will sign a memorandum of agreement (MOA), with the understanding that they may be randomized into an intervention or control condition. The MOA outlines the responsibilities of the research team and the participating sites and a list of benefits of participation. Eligibility criteria for Head Start centers will be: a) students are predominantly American Indian or Hispanic; b) a minimum of 20 3-year olds are enrolled each year; and c) the center retains at least 80% of its students for two years. Head Start children and their families will be recruited for CHILE upon their enrollment in the participating Head Start centers. For Head Start children to be eligible for the study, they must be enrolled in one of the participating Head Start centers, be 3 years old at baseline, and have an active consent form completed by their parent or legal guardian. The primary caregiver for each participating Head Start student will also participate in the study. In addition, Head Start teachers, aides, and food service workers/cooks affiliated with the 16 Head Start centers will be involved in the study, through participation in intervention training and implementation, periodic interviews and/or focus groups, and completion of written logs. In intervention Head Start communities, grocery store managers and owners, as well as the Head Start teachers, aides, and food service workers/cooks, will be involved in the intervention.

Formative assessment will take place during the first six months of the study to ensure that the intervention will meet the needs, context, and the daily realities of working in Head Start centers and communities in rural New Mexico. Similar to the principles set by the UNM PRC in other community-based participatory research efforts, and consistent with the aims of this study, the formative assessment will examine Head Start barriers and resources, and identify with Head Start staff the opportunities for integrating physical activity and nutrition into the curricula, food service, and general Head Start environment. The information gathered during this period will be used to adapt and/or design developmentally-appropriate, organizationally-feasible physical activity and nutrition interventions for the schools. Priority will be given to intervention components that have proven to be feasible in other studies. After developing and signing an MOA with each intervention and control Head Start center that outlines research study aims and roles and responsibilities, study staff will use a modified version of the Environmental Checklist developed for Pathways to identify potential environmental foci for change.

Observations of Head Start students during recess, before school, at lunch, and at other "open" times will be conducted by members of the research team at Head Start centers to gain information about their level and intensity of physical activity during the school day, as well as to identify locations used for physical activity.

Finally, during the formative assessment phase, height and weight data will be collected for current Head Start students (not study participants), so that Head Start centers can be grouped by median BMI percentile values for randomization.

Following the formative assessment, Head Start centers will be randomly assigned to the intervention or control condition. To ensure that the baseline average BMI percentile will be similar in control and intervention groups, Head Start centers will be assigned by a stratified randomization process. We expect 10 predominantly Hispanic Head Starts and 6 predominantly American Indian Head Starts. Pre-intervention baseline measurements made at each Head Start center will be used to stratify Head Start centers in each ethnic subpopulation into lower and upper BMI percentile strata. Random allocation will be used to assign intervention status in strata defined by BMI and ethnicity.

Once the intervention Head Start centers have been determined, intervention planning will be conducted with these centers. The interventionists will coordinate efforts to integrate Head Start staff, community leaders, health providers, and grocery store managers and owners in the strategic planning process for the intervention. The purpose of this phase is to establish a collaborative relationship with study participants and to ensure that the intervention materials and curriculum reflect the cultural context of each community. While the study team has collectively conducted research in many of the proposed communities, it is essential to establish a participatory framework that can be sustained throughout the duration of the study and beyond.

Strategies will include: hands-on food preparation and taste-testing of fruits, vegetables, and whole grain foods; and story telling, poems, songs, games, crafts, and/or puppets to reinforce familiar and introduce new fruits, vegetables and whole grain foods. Materials will be sent home with students so that the intervention activities can be reinforced with the families.

Head Start staff play a critical role in the intervention. They will receive in-service training on a quarterly basis designed to prepare and support them in implementing the classroom curriculum. We anticipate that frequent training for shorter periods of time than Pathways teacher training will keep the intervention fresh and the content more manageable. Topics will include the importance of obesity prevention, the role of fruits, vegetables, and whole grains in maintaining weight and preventing obesity, the role of physical activity in maintaining weight and preventing obesity, developmentally appropriate physical activity, and strategies for limiting television viewing and other screen time. Much of the training will be hands-on and experiential learning, like many of the activities they will be conducting in the classroom. We will also work with the Head Start program staff to determine the feasibility of our training sessions contributing to the credentialing process for Head Start teachers and other staff.

We plan to use a training program for the Head Start cooks of the intervention schools similar to the successful school food service training program used with the Pathways intervention. The focus will be on preparing and serving meals that meet the recently revised Dietary Guidelines for Americans (2005). Annual training sessions will be reinforced by monthly visits to each intervention Head Start school. Our experience with the Pathways program suggests that federally mandated nutrition programs (such as the National School Lunch and School Breakfast Programs) are not necessarily followed precisely at individual sites, so we will emphasize the Dietary Guidelines and reinforce the NSLP and SBP requirements during training sessions and follow-up visits to the centers. As with schools participating in the Pathways program, we anticipate the training sessions and visits will be met with enthusiasm.

To engage family support and involvement in CHILE, the intervention will include both home- and Head Start-based activities for families. The home-based component will include activities that parents can do with their children at home, such as preparing healthful snacks, taking a walk, and playing active games together. These activities will be introduced at the Family Events, which will be held four times each year, and will be re-enforced with take home material. Families will be asked to limit television viewing and other screen time to 2 hours or less per day. This too will be introduced and re-enforced at Family Events. Family Events will include such activities as hands-on food preparation and taste-testing of fruits, vegetables, and whole grain foods, label reading, grocery store field trips, "Ask the Doctor" (a special one-on-one interaction with a local participating health care provider), and booths demonstrating concepts and content children are learning in the classroom.

ELIGIBILITY:
Inclusion Criteria:

* 3 years of age of beginning of intervention for each cohort (2)
* enrolled in participating Head Start
* informed consent signed by parent or legal guardian

Exclusion Criteria:

* 4 years of age or more at beginning of intervention for each cohort (2)
* not enrolled in a participating Head Start
* informed consent not provided

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 980 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Increase physical activity | 2010
Increase the intake of fiber | 2010
Decrease fat intake | 2010
Decrease television and other screen time | 2010
Decrease obesity | 2010

SECONDARY OUTCOMES:
Changes in Head Start and community policy in regards to physical activity | 2010
Changes in Head Start and community policy in regards to school food service | 2010
Changes in Head Start and community policy in regards to school snacks | 2010
Changes in Head Start and community policy in regards to availability of healthful options | 2010
Examine the role of community leaders in raising awareness of obesity prevention | 2010
Examine the role of community leaders in creating a supportive environment for the prevention of obesity | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Sally M Davis, Ph.D., Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Morshed AB, Davis SM, Keane PC, Myers OB, Mishra SI. The Impact of the CHILE Intervention on the Food Served in Head Start Centers in Rural New Mexico. J Sch Health. 2016 Jun;86(6):414-23. doi: 10.1111/josh.12393. PMID 27122141
- [Derived] Cruz TH, Davis SM, Myers OB, O'Donald ER, Sanders SG, Sheche JN. Effects of an Obesity Prevention Intervention on Physical Activity Among Preschool Children: The CHILE Study. Health Promot Pract. 2016 Sep;17(5):693-701. doi: 10.1177/1524839916629974. Epub 2016 Apr 18. PMID 27091603
- [Derived] Cruz TH, Davis SM, FitzGerald CA, Canaca GF, Keane PC. Engagement, recruitment, and retention in a trans-community, randomized controlled trial for the prevention of obesity in rural American Indian and Hispanic children. J Prim Prev. 2014 Jun;35(3):135-49. doi: 10.1007/s10935-014-0340-9. PMID 24549525